CLINICAL TRIAL: NCT00456612
Title: Phase I/II Study of Fractionated CyberKnife Stereotactic Radiosurgery for High Grade Gliomas in Elderly Patients With Poor Performance Status
Brief Title: Radiosurgery for Glioblastoma Multiforme
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Anand Mahadevan, Radiation Oncologist, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006P-000464
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyberknife (Other): Radiosurgery to enhancing high grade glioma in 5 fractions with escalating doses.
  Interventions: Procedure: CyberKnife

INTERVENTIONS:
Procedure: CyberKnife — Radiosurgery to enhancing high grade glioma in 5 fractions with escalating doses.

SUMMARY:
Conventional radiation for 6 weeks is not well tolerated by the elderly. Shorter courses (over 3-5 weeks) of radiation have been shown to be equivalent in outcome the elderly- particularly in patients who are generally in poor performance status (KPS<70). Fractionated Cyberknife Radiosurgery can deliver equivalent doses in 5 treatments providing the same tumor control in a much shorter and tolerable schedule improving their quality of their short life.

To assess the tolerability of Cyberknife Radiosurgery for High Grade Gliomas in Elderly with poor performance status.

Secondary:

Assessment of local control rate, progression free survival, overall survival, quality of life and toxicity and steroid dependence in this population with this regime.

DETAILED DESCRIPTION:
Conventional radiation for 6 weeks is not well tolerated by the elderly. Shorter courses (over 3-5 weeks) of radiation have been shown to be equivalent in outcome the elderly- particularly in patients who are generally in poor performance status (KPS<70). Fractionated Cyberknife Radiosurgery can deliver equivalent doses in 5 treatments providing the same tumor control in a much shorter and tolerable schedule improving their quality of their short life.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed newly diagnosed glioblastoma multiforme or Anaplastic Glioma (WHO Grade III) by surgical excision or biopsy.
2. Patient must recover from the effects of surgery, post-operative infection, or other complications.
3. Therapy should start within 5 weeks of surgery
4. Must have an estimated survival of > 8 weeks.
5. KPS < 70.
6. Age > 65 years.
7. Must have a pre- and post operative contrast enhanced MRI scans
8. Laboratory values within the following limits: ANC (absolute neutrophil count) >/= 1500 cell/ul Platelets >/= 100x 10(3)/ul, Hemoglobin >/= 9g/dl, Serum Creatinine ≤ 1.5mg/dl., Serum total Bilirubin </= 1.5 x upper limit of normal (ULN), SGOT/SGPT </= 2.5x ULN, Albumin >/= 3g/dl.

   -

Exclusion Criteria:

1. Histology grade less than Anaplastic Glioma ( WHO Grade III).
2. Recurrent malignant glioma.
3. Tumor involving the Brain stem.
4. Any detected tumor foci beyond the cranial vault.
5. Major medical or psychiatric illness, which in the investigator's opinion will prevent administration or completion of the protocol therapy.
6. Prior malignancies, except for non-melanomatous skin cancers, or carcinoma in situ of uterus, cervix or bladder, unless disease free for > 5 years.
7. Prior chemotherapy for the current disease.

   -

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Mahadevan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyberknife
Started | 4
Completed | 1
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Single arm Phase II Study
Arm/Group | Single Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: The Percent Progression -Free Survival at 6 Months Will be Tabulated
Time Frame: 6 months
Arm/Group | Cyberknife
Number analyzed (Participants) | 0

2. Secondary Outcome: Response, Median Time to Tumor Progression,Overall Survival, Percent Overall Survival at 1 Year Will be Tabulated.
Time Frame: 1year
Reporting Status: Not Posted

3. Primary Outcome: Progression Free Survival
Time Frame: consent to prgression or death
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Single Arm Study: Single arm Phase II Study
Arm/Group | Single Arm Study
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Early termination due to difficulty in recruitment and retaining due to extremely bad prognosis of disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No